CLINICAL TRIAL: NCT04045639
Title: A Randomised Controlled Trial for the Identification of Undiagnosed Atrial Fibrillation Patients Using a Machine Learning Risk Prediction Algorithm and Diagnostic Test
Brief Title: A Study to Assess the Effectiveness of an Atrial Fibrillation (AF) Risk Prediction Algorithm and Diagnostic Test in Identifying Patients With AF.
Acronym: PULsE AI
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-703
Record Dates: First submitted 2019-07-23; First posted 2019-08-05 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention arm: The AF risk prediction algorithm will be run on patient records within the Egton Medical Information Systems (EMIS) data base, in order to identify patients at risk of developing AF
- Control arm: Patients may be diagnosed with AF through routine clinical practice only

SUMMARY:
This is a trial to assess the effectiveness of an atrial fibrillation (AF) risk prediction algorithm and diagnostic test for the identification of patients with atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

Practice inclusion criteria for the trial are as follows;

* GP Practices within National Institute for Healthcare Research (NIHR) Clinical Research Network: West Midlands (CRN: WM) CRN: WM
* GP Practices using EMIS as their electronic medical record system of choice. Patient inclusion criteria for the trial are as follows;
* Patients registered at a participating practice, aged ≥30 years and without an AF diagnosis.
* Patients with a valid index date (see Section 3.3) Participant inclusion criteria for participation in the intervention arm are;
* As above, and who have provided written consent to: attend a research clinic, AF diagnosis check using a 12-lead ECG, and for access to medical records Participant inclusion criteria for participation in further AF remote diagnosis with an AliveCor Heart Monitor are;
* As above, and those with a negative or indeterminant ECG
* As above, and those with access to a smartphone

Exclusion criteria:

* Patients <30 years
* Patients with an existing diagnosis of AF
* Patients for whom the healthcare professional feels the study is unsuitable

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is anticipated that approximately 18,000 patient records will be included in the trial.
  It is anticipated that approximately 1,200 undiagnosed patients would be invited for AF diagnosis across all study sites.30 years is taken as the minimum age entry criteria as the algorithm was built on information from patients >30 years where AF becomes more prevalent.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with diagnosed Atrial Fibrillation during the research window in control and intervention arms | From the first collection of patient medical records at the beginning of the trial to the last collection of patient records following the intervention at the end of the trial (Up to 6 months)
  Prevalence of AF in the research window assessed

SECONDARY OUTCOMES:
Expected healthcare resource utilisation (Annual maintenance costs related to health states (informed by the primary endpoint), and daily treatment costs (including monitoring)) | Up to 6 months
Quality-adjusted life years (QALYs) | Up to 6 months
Life years (LYs) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United Kingdom (6):
  - Local Institution, Ludlow
  - Local Institution, Royal Leamington Spa
  - Local Institution, Shropshire
  - Local Institution, Warkwickshire
  - Local Institution, Wolverhampton
  - Local Institution, Worcester

REFERENCES:
- [Derived] Hill NR, Arden C, Beresford-Hulme L, Camm AJ, Clifton D, Davies DW, Farooqui U, Gordon J, Groves L, Hurst M, Lawton S, Lister S, Mallen C, Martin AC, McEwan P, Pollock KG, Rogers J, Sandler B, Sugrue DM, Cohen AT. Identification of undiagnosed atrial fibrillation patients using a machine learning risk prediction algorithm and diagnostic testing (PULsE-AI): Study protocol for a randomised controlled trial. Contemp Clin Trials. 2020 Dec;99:106191. doi: 10.1016/j.cct.2020.106191. Epub 2020 Oct 19. PMID 33091585
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm